CLINICAL TRIAL: NCT06916273
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of PA9159 Inhalation Aerosol in Healthy Adult Subjects in China
Brief Title: Safety, Tolerability, and Pharmacokinetics of PA9159 Inhalation Aerosol in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA9159AS-101
Record Dates: First submitted 2025-03-12; First posted 2025-04-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Arm 1-4, the treatment is given once for one day, with escalation doses of 60 μg, 120 μg, 240 μg, 300 μg. For each dose group, 6, 8, 8 and 8 healthy subjects will be randomly assigned in a 2:1, 3:1, 3:1 and 3:1 ratio respectively to receive the test drug PA9159 inhalation aerosol or placebo. Arm 5, PA9159 at the escalation dose of 120 μg is given twice a day for 7 days. 10 health subjects will be enrolled for this dose group, randomized proportionally at 4:1 ratio to receive either the investigational product PA9159 Inhalation aerosol or placebo , with a total of 40 subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PA9159 60 μg single dose and placebo (Experimental): Six subjects will be randomly assigned at a 2:1 ratio to receive either single dose of 60 μg PA9159 or placebo. Before escalating to the next dose level, all available clinical and laboratory safety data will be reviewed.
  Interventions: Drug: PA9159 Inhalation aerosol, 60 μg one day treatment; Drug: Placebo, the same Inhalation aerosol solution without PA9159 active ingredient
- PA9159 120 μg single dose and placebo (Experimental): Eight subjects will be randomly assigned in a 3:1 ratio to receive either single dose of 120 μg PA9159 or placebo. Before escalating to the next dose level, all available clinical and laboratory safety data will be reviewed.
  Interventions: Drug: PA9159 Inhalation aerosol, 120 μg one day treatment; Drug: Placebo, the same Inhalation aerosol solution without PA9159 active ingredient
- PA9159 240 μg single dose and placebo (Experimental): Eight subjects will be randomly assigned in a 3:1 ratio to receive either single dose of 240 μg PA9159 or placebo. Before escalating to the next dose level, all available clinical and laboratory safety data will be reviewed.
  Interventions: Drug: PA9159 Inhalation aerosol, 240 μg one day treatment; Drug: Placebo, the same Inhalation aerosol solution without PA9159 active ingredient
- PA9159 300 μg single dose and placebo (Experimental): Eight subjects will be randomly assigned in a 3:1 ratio to receive either single dose of 300 μg PA9159 or placebo. all available clinical and laboratory safety data will be reviewed.
  Interventions: Drug: PA9159 Inhalation aerosol, 300 μg one day treatment; Drug: Placebo, the same Inhalation aerosol solution without PA9159 active ingredient
- PA9159 120 μg repeated doses and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either 120 μg PA9159 or placebo twice a day for 7 days. all available clinical and laboratory safety data will be reviewed.
  Interventions: Drug: PA9159 Inhalation aerosol, 120 μg 7-day treatment; Drug: Placebo, the same Inhalation aerosol solution without PA9159 active ingredient

INTERVENTIONS:
Drug: PA9159 Inhalation aerosol, 60 μg one day treatment — single dose of PA9159 (60 μg/inhaler spray) is administered by inhalation through an inhaler via the mouth, with 2 puffs.
  Arms: PA9159 60 μg single dose and placebo
Drug: PA9159 Inhalation aerosol, 120 μg one day treatment — single dose of PA9159 (120 μg/inhaler spray) is administered by inhalation through an inhaler via the mouth, with 4 puffs.
  Arms: PA9159 120 μg single dose and placebo
Drug: PA9159 Inhalation aerosol, 240 μg one day treatment — single dose of PA9159 (240 μg/inhaler spray) is administered by inhalation through an inhaler via the mouth, with 8 puffs.
  Arms: PA9159 240 μg single dose and placebo
Drug: PA9159 Inhalation aerosol, 300 μg one day treatment — single dose of PA9159 (300 μg/inhaler spray) is administered by inhalation through an inhaler via the mouth, with 10 puffs.
  Arms: PA9159 300 μg single dose and placebo
Drug: PA9159 Inhalation aerosol, 120 μg 7-day treatment — Repeated doses of PA9159 (120 μg/inhaler spray) i is administered by inhalation through an inhaler via the mouth, with 4 puffs, twice a day.
  Arms: PA9159 120 μg repeated doses and placebo
Drug: Placebo, the same Inhalation aerosol solution without PA9159 active ingredient — Placebo is delivered via the mouth through an inhaler with the same volume as the corresponding PA9159 dose group

SUMMARY:
PA9159 is a highly potent novel corticosteroid. The purpose of this study is to exam the safety, tolerability, and pharmacokinetics of single and repeat dosing of Inhalation aerosol PA9159, to establish maximum tolerated dose in healthy chinese adult

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled dose escalation phase 1 trial, including single dose and 7-day repeat doses of PA9159 Inhalation aerosol. In the first part of the study, the treatment is given once for one day, with escalation doses of 60 μg, 120 μg, 240 μg, 300 μg. 30 health subjects will be enrolled for this part. In the second part of the study, PA9159 at the escalation dose of 120 μg is given twice a day for 7 days. 10 health subjects will be enrolled for this group, randomized proportionally at 4:1 ratio to receive either the investigational product PA9159 Inhalation aerosol or placebo , with a total of 40 subjects for this two-part study. Subjects will be evaluated for the safety, tolerability and pharmacokinetics of PA9159 Inhalation aerosol.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 65 years (including upper and lower limits);
* Male body weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) between 19 and 26 kg/m2 (including cut-off values);
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Those who cannot use the nebulizer correctly, cannot tolerate nebulized inhalation administration or have failed the training for inhalation administration;
* Those with special dietary requirements and cannot follow the unified diet;
* Those with a history of chronic diseases such as cardiovascular, digestive, endocrine, hematological, immune, and nervous system diseases; those with chronic diseases of the oral, pharyngeal, and respiratory systems; those with chronic diseases of the oral, pharyngeal, and respiratory systems at the time of screening; those with a history of recurrent (defined as more than 1 episode) or disseminated herpes zoster, repeated infection, tuberculosis infection, glaucoma, or cataract;
* Those who are allergic to the study drug or any component of the study drug, or have an allergic constitution (referring to an allergic constitution to more than two drugs and foods);
* Those whose vital signs, physical examination, laboratory tests, chest X-ray examination, 12-lead electrocardiogram examination, pulmonary ventilation function examination, etc. at the screening period are judged abnormal and have clinical significance;
* Those with positive tests for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), Treponema pallidum antibody (Syphilis TP), human immunodeficiency virus (HIV Ag/Ab);
* Those with FEV1 ≤ 80% of predicted value or FVC ≤ 80% of predicted value at the screening period;
* Those who frequently drink alcohol within 3 months before screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer with 5% alcohol content or 45 mL of spirits with 40% alcohol content or 150 mL of wine with 12% alcohol content) or those with positive alcohol breath test at the screening period or those who cannot stop alcohol intake during the study period;
* Those with a smoking history of more than 10 years and smokers within 3 months before screening, or those who cannot stop using any tobacco products during the trial, or those with positive nicotine detection at the baseline period.
* Those who have a history of drug abuse or drug use within the past two years, or those whose urine screening for drug abuse is positive;
* Those who have taken any drugs (prescription drugs, over-the-counter drugs, Chinese herbal medicines, vaccines) or health supplements within the two weeks prior to screening or during the screening period;
* Those who have used any preparations containing glucocorticoid components or any drugs that affect the activity of CYP3A4 enzymes (such as ritonavir or ketoconazole, etc., as detailed in Appendix 5) within the 30 days prior to screening or during the screening period;
* Those who have consumed beverages or foods containing grapefruit, dragon fruit, mango, pomelo, pomegranate, papaya, or rambutan within 14 days prior to screening or during the screening period, or those who do not agree to stop consuming the above foods during the trial period;
* Those who have consumed any foods or beverages rich in caffeine, xanthine within 48 hours before the first use of the study drug (coffee, tea, cola, chocolate, seafood, animal liver, etc.), or those who do not agree to stop consuming the above foods during the trial period;
* Those who have donated blood or suffered significant blood loss within 90 days prior to screening or during the screening period (≥ 400 mL, except during the menstrual period of women) or have received blood products or undergone blood transfusion;
* Those who have participated in other clinical trials within 90 days prior to screening and have used the study product;
* Those who have undergone respiratory surgery in the past, or those who have undergone major surgery within 3 months prior to screening (judged by the investigator based on the previous medical history), suffered major trauma or planned to undergo surgery during the trial period;
* Those who have difficulty in venous blood collection, or have a known history of multiple fainting or hematemesis;
* Female subjects who have tested positive for pregnancy detection or are in lactation during the screening period or baseline period;
* Subjects who, in the opinion of the investigator, have other conditions that are not suitable for participating in the trial or who cannot participate in the trial due to their own reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events (AEs) | within 48 hours after last treatment
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Number of subjects having abnormal hematology laboratory parameters | within 48 hours after last treatment
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal clinical chemistry parameters | within 48 hours after last treatment
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal values for urinalysis | within 24 hours after last treatment
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Systolic and diastolic blood pressure | within 48 hours after last treatment
  Vital sign-Systolic and diastolic blood pressure
ECG parameter-QTc interval | up to 24 hours after last treatment
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically calculates the QTc intervals
Body temperature | within 48 hours after last treatment
  Vital sign-Body temperature
Pulse rate | within 48 hours after last treatment
  Vital sign-Pulse rate
ECG parameter-PR interval | up to 24 hours after last treatment
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures PR intervals
ECG parameter-QRS duration | up to 24 hours after last treatment
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures QRS duration

SECONDARY OUTCOMES:
Serum cortisol levels | From pre-dose until 24 hours post-dose
  Monitor the concentration changes of serum cortisol before and after PA9159 administration.
Pharmacokinetics of single dose and repeat doses of inhalation aerosol PA9159 | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects)5, 10, 15, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter (Cmax）
Pharmacokinetics of single dose and repeat doses of inhalation aerosol PA9159 | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects)5, 10, 15, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter (Tmax)
Pharmacokinetics of single dose and repeat doses of inhalation aerosol PA9159 | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects)5, 10, 15, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter (AUC)
Pharmacokinetics of single dose and repeat doses of inhalation aerosol PA9159 | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects)5, 10, 15, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Wen, phD, Principal Investigator — The First Affiliated Hospital of Nanchang University; Xiaohua Cheng, Master, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No